CLINICAL TRIAL: NCT02671825
Title: A Phase 1 Single Center, Single Group, 7-way Crossover Pilot Pharmacokinetic Study to Evaluate the Disposition of Active Component Following Single Inhaled Doses of Five Formulations of PUR0200 Compared to Reference Product in Healthy Adult Subjects
Brief Title: A PK Study to Evaluate PUR0200 and a Reference Product in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 601-0012P
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- PUR0217a (Experimental): PUR0200 formulation 1
  Interventions: Drug: PUR0200
- PUR0228a (Experimental): PUR0200 formulation 2
  Interventions: Drug: PUR0200
- PUR0228b (Experimental): PUR0200 formulation 3
  Interventions: Drug: PUR0200
- PUR0228c (Experimental): PUR0200 formulation 4
  Interventions: Drug: PUR0200
- PUR0230c (Experimental): PUR0200 formulation 5
  Interventions: Drug: PUR0200
- Reference Product 1 (Active Comparator): Reference Product formulation with active charcoal
  Interventions: Drug: Reference Product
- Reference Product 2 (Active Comparator): Reference Product without active charcoal
  Interventions: Drug: Reference Product

INTERVENTIONS:
Drug: PUR0200 — PUR0200 dry powder inhalation
  Arms: PUR0217a; PUR0228a; PUR0228b; PUR0228c; PUR0230c
Drug: Reference Product — Dry Powder Inhalation Reference Product
  Arms: Reference Product 1; Reference Product 2

SUMMARY:
The purpose of this study is to compare drug blood levels of multiple formulations of inhaled PUR0200 to each other and to the reference product with and without oral charcoal.

DETAILED DESCRIPTION:
The purpose of this study is to compare 5 different formulations of PUR0200 to the reference product. All formulations will be inhaled. In 6 of the 7 study periods either PUR0200 or the reference product will be inhaled under fasting conditions without oral charcoal. In the 7th study period, half of the subjects will receive reference with oral charcoal and the other half will receive reference product without oral charcoal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject
* Age between 18 and 50 (inclusive) years
* Non-smokers or ex-smokers (stopped at least 6 months ago)
* FEV1 ≥80% of the predicted value
* Completion of 3 training inhalations

Exclusion Criteria:

* Pregnant and/or nursing women. Positive pregnancy test at entry visit or on hospitalization day 0 of each study period.
* fertile women without reliable contraception
* participation in ANY research study within 3 months prior to entry visit, or simultaneous participation in another clinical study
* blood donation or blood loss within last 3 months
* treatment with ANY investigational study drug (i.e. drug not yet approved) in the last 3 months before entry visit
* intake or administration of any prescribed systemic or topical medication including over the counter (OTC) medication or natural food supplements (e.g. vitamins, garlic, or ginger capsules) within 2 weeks before entry visit
* current or history of drug abuse within 5 years before entry visit
* alcohol abuse
* regular consumption of beverages or food containing methylxanthines (i.e. coffee, tea, cola, caffeine containing sodas, chocolate) equivalent to more than 500 mg methylxanthines* per day
* presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, hematological, gastrointestinal, neurological, psychiatric or other diseases
* major surgery of the gastrointestinal tract except for appendectomy, or any pulmonary surgery
* clinically significant illness (including upper or lower respiratory infection and/or candidiasis of the mouth and throat) within 4 weeks before entry visit
* any acute or chronic disease which might interfere with inhalation, absorption, distribution, metabolism or excretion of the drug special diet due to any reason, e.g. vegetarians
* positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies
* excessive physical activity (more than 4 times per week for more than 90 minutes) within the last 6 months and during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To assess PK parameter area under the plasma concentration versus time curve (AUC) of 5 formulations of PUR0200 compared to Reference Product | 8 hours
To assess PK parameter Peak Plasma Concentration (Cmax) of 5 formulations of PUR0200 compared to Reference Product | 8 hours

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events | 8 weeks
  self-reported and investigator-assessed adverse events, vital signs, and laboratory safety examinations
Comparison of PK parameters (AUC and Cmax) in subjects dosed with Reference product after ingesting charcoal and without charcoal to assess oral vs inhalation exposure of drug | 8 hours
Comparison of PK parameters (AUC and Cmax) in subjects dosed with Reference product in 2 separate periods to assess the intra-subject variability of inhalation exposure to Reference product | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Kirkov, MD, Principal Investigator — Tokuda Hospital; David Hava, PhD, Study Director — Pulmatrix Inc.
Locations (1):
- Tokuda Hospital, Sofia, Bulgaria